CLINICAL TRIAL: NCT04075838
Title: The Development and Efficacy of a Recovery Group for People With Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-ER-106-245
Record Dates: First submitted 2019-07-16; First posted 2019-09-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-07

CONDITIONS: Mental Illness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recovery group (Other): The researchers designed a recovery group suited to Taiwanese with mental illness, according to content of the PTR (Ridgway et al., 2002) and recovery-related literature (Davidson et al., 2005; Ridgway, 2001). The group gathered for a one-hour session once a week for 18 weeks.
  Interventions: Other: Recovery group

INTERVENTIONS:
Other: Recovery group — The researchers designed a recovery group suited to Taiwanese with mental illness, according to content of the PTR (Ridgway et al., 2002) and recovery-related literature (Davidson et al., 2005; Ridgway, 2001)

SUMMARY:
Recovery-oriented approach has been promoted in psychiatric rehabilitation in recent years. This approach emphasizes that people with mental illness can live a hopeful life even though the symptoms still exist. However, few recovery-oriented programs are available in Taiwan. This study aimed to develop of a recovery-oriented program for people with mental illness and investigate its feasibility.

DETAILED DESCRIPTION:
The study participants with mental illness were from a community mental health center in the south of Taiwan. The recovery-oriented program was conducted by a group leader, a senior occupational therapist, with one supervisor and one observer. The program was designed based on Pathways to Recovery, a self-help book published by University of Kansas. Participants attended a 1-hour class per week. The teaching methods included didactic presentation, peer exchange, group discussion, and practice. The group leader, supervisor, and observer reviewed the content and participants' performance after each class and made content adjustments if needed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mental illness

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
Stages of Recovery Scale：Change from Baseline at 10 weeks and 18 weeks | baseline, 10 weeks, 18 weeks
  The scale consists of 45 items, with six subscales: the sense of hope, disability management/taking responsibility, regaining autonomy, social functioning/role performance, overall well-being, and willingness to help. It has good internal consistency and proper construct validity. The SRS utilizes a 4-point rating scale: never (0), seldom (1), sometimes (2), and often (3). Higher scores indicate better recovery. The developers also provide the cutoff scores for four recovery stages: Stage 1 (overwhelmed by the disability), 0-57; Stage 2 (struggling with disability), 58-90; Stage 3 (living with disability), 91-119; and Stage 4 (living beyond disability), 120-135.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Yen-Ching, Study Chair — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No